CLINICAL TRIAL: NCT06114680
Title: Evaluation of the CochSyn Test Prototype to Measure Cochlear Synaptopathy
Acronym: EarDiTech
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Delay in recruitment and funding exhausted
Sponsor: University Ghent (Other)
Collaborators: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ONZ-2023-0258
Record Dates: First submitted 2023-09-29; First posted 2023-11-02 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-04

CONDITIONS: Hearing Loss, Sensorineural; Cochlear Synaptopathy; Cochlear Hearing Loss
MeSH Terms: conditions — Hearing Loss, Sensorineural; Hearing Loss, Hidden

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Session 1 - test group (self-reported hearing difficulties) (Other): 143 (130 + 10% potential drop-outs) subjects with self-reported hearing difficulties according to the HHIE-s questionnaire (score of >4)
  Interventions: Device: CochSyn test prototype; Device: Universal Smart Box (USB)
- Session 1 - control goup (no self-reported hearing difficulties) (Other): 66 (60 + 10% potential drop-outs) subjects with no self-reported hearing difficulties according to HHIE-s questionnaire (score of ≤4)
  Interventions: Device: CochSyn test prototype; Device: Universal Smart Box (USB)
- Session 2 (self-reported hearing difficulties) (Other): 66 (60 + 10% potential drop-outs) subjects who participated in session 1 - test group
  Interventions: Device: CochSyn test prototype

INTERVENTIONS:
Device: CochSyn test prototype — The CochSyn test prototype is intended for use in the evaluation of hearing-related disorders in adults using auditory evoked potentials. The CochSyn test prototype records biopotential waveforms that can be used for hearing screening and diagnostic applications.
Device: Universal Smart Box (USB) — Commercially available EEG system intended for use in the diagnosis of hearing related disorders, hearing threshold detection, and other conditions that may affect the responses to auditory, tactile, or visual stimuli. The USB Box hardware and accompanying software programs can be used with patients of all ages. It is intended for use by trained personnel in a hospital, nursery, clinic, audiologist's office, or other appropriate setting.
  Arms: Session 1 - control goup (no self-reported hearing difficulties); Session 1 - test group (self-reported hearing difficulties)

SUMMARY:
This study investigates a newly developed test, The CochSyn test that can quantify cochlear synaptopathy (CS) (a new type of sensorineural hearing loss (SNHL)) earlier than the current golden standard pure-tone audiogram.This newly developed test is based on auditory evoked brain potentials. A hardware prototype (the Cochsyn test prototype) was developed to use the Cochsyn test in clinical practice. Additionally a CS-based sound-processing algorithm (CoNNear) that is designed to improve speech intelligibility in subjects that are identified to have CS, will be investigated in this study.

DETAILED DESCRIPTION:
Cochlear synaptopathy is a new type of sensorineural hearing loss (SNHL) and is related to ageing, noise exposure and ototoxicity. There is currently no diagnostic test of CS on the market, whereas CS is an important form of SNHL. CS occurs before the golden standard clinical hearing test (pure- tone audiogram in which participants raise their hand when hearing tones of different frequencies and the threshold of hearing is determined), shows any signs of hearing damage.

The investigators have developed a test, the CochSyn test that may quantify SNHL earlier than the audiogram. The newly developed test is based on auditory evoked potentials. This is a method in which an auditory stimulus is presented, and encephalogram (EEG) electrodes capture the sound-evoked brain potentials. The most popular auditory evoked potential metric to diagnose sensorineural hearing loss (SNHL) is the auditory brainstem response (ABR). The first animal research studies on CS confirmed that the ABR wave-I amplitude is a sensitive marker of CS when the inflicted hearing damage is well-controlled and specific. Even though it can be assumed that the ABR wave-I amplitude will also be sensitive to CS in humans, it may not be a differential marker for it, and hence other candidate auditory evoked potential markers for CS have been investigated in recent studies. In particular, the envelope-following-response (EFR), has also been shown to be specific to CS in animal research studies.

EFRs are recorded using the standard ABR electrode montage but use another type of stimulus. Based on model simulations and a recent study in which the investigators compared candidate EFR markers for use in human studies , the investigators have developed a new stimulus for EFRs that uses both a different type of modulator waveform and a different analysis method than was adopted earlier.

In this trial, the investigators wish to test the performance of the new method (the CochSyn test) in listeners with or without self-reported hearing difficulties using a newly developed hardware prototype (the CochSyn test prototype), dedicated for the CochSyn-test in clinical practice. The assessment also includes the testing of a CS-based sound-processing algorithm (CoNNear) that is designed to improve speech intelligibility in subjects that are identified to have CS, based on our CochSyn test.

To this end, the investigators will first assess whether our CochSyn test prototype is equally good at capturing the standard ABR waveform as a comparator device available on the market (the Intelligent Hearing Systems Universal Smart Box). The investigators will also test which stimulation characteristics and electrode configurations for the CochSyn test are best able to quantify individual differences in standard objective hearing tests (audiogram, otoacoustic emission, speech reception thresholds) and subjective hearing complaints (validated HHIE-s questionnaire).

ELIGIBILITY:
Inclusion Criteria:

Session 1

Test group

* 18 - 87 years old
* Flemish/Dutch as native language
* Ability to fill out a questionnaire and to perform a speech intelligibility test
* Self-reported hearing difficulties according to HHIE-s questionnaire (score of >4)
* Normal audiogram (for age group 18-77): audiometric thresholds up to 4 kHz ≤ 20 dB HL and for 6 kHz ≤ 40 dB HL in at least 1 ear OR impaired audiogram (for age group 18-87): audiometric thresholds between 20.1 and 64.9 dB HL pure tone average at 0.5, 1, 2, and 4 kHz in at least 1 ear (=Mild to moderately severe hearing loss according to the recommendation by the Global Burden of Disease Expert Group on Hearing Loss)

Control group

* 18 - 77 years old
* Flemish/Dutch as native language
* Ability to fill out a questionnaire and to perform a speech intelligibility test
* No self-reported hearing difficulties according to HHIE-s questionnaire (score of ≤4)
* Normal audiogram: audiometric thresholds up to 4 kHz ≤ 20 dB HL and for 6 kHz ≤ 40 dB HL in at least 1 ear

Session 2

* Participation in session 1 in the test group
* 18 - 77 years old
* EFR magnitude at 4 kHz with Snap electrode in session 1 reduced by 30-100% compared to average EFR magnitude of age group 18-27 of control group (session 1)

Exclusion Criteria:

Applicable for both sessions:

* Pregnant woman
* Breastfeeding woman

Applicable for both sessions and the ear which fulfils the inclusion criteria:

* Chronic (longer than 6 months) permanent tinnitus
* Hearing loss due to a genetic condition, a middle ear condition, or surgery
* Congenital hearing loss
* Blocked ear canal

Ages: 18 Years to 87 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 179 (Actual)
Dates: Start 2023-11-13 (Actual); Primary Completion 2025-12-23 (Actual); Study Completion 2025-12-23 (Actual)

PRIMARY OUTCOMES:
Quality of Cochsyn test prototype | end of session 1, after 3 hours
  The difference in terms of wave amplitudes of a standard clinical auditory brainstem response (ABR) recorded with the commercially available USB device and with the CochSyn test prototype during session 1.
Sensitivity CochSyn test prototype | end of session 1, after 3 hours
  The difference in sensitivity (i.e., standard deviation/range) between the ABR wave-I amplitude and the EFR magnitude as measured on the CochSyn test prototype with Snap electrodes in session 1.

SECONDARY OUTCOMES:
Usability CochSyn test prototype | end of session 1, after 3 hours
  Written feedback in form of a questionnaire of the test administrator on the usability of the test system for the measurements performed with the CochSyn test prototype during session 1.
Performance CochSyn test prototype | end of session 1, after 3 hours
  The difference between the EFR magnitudes obtained with the CochSyn test prototype + cEEGrid electrodes and those obtained with the CochSyn test prototype + Snap electrodes measured for different stimulus carriers during session 1.
Reliability Cochsyn test prototype | end of session 2, after 2 hours
  The difference between the EFR magnitudes during session 1 and session 2 (test/re-test). This concerns the recordings made with the CochSyn test prototype + cEEGrid and with the CochSyn test prototype + Snap electrodes.
Sensitivity related to stimulus changes | end of session 1, after 3 hours
  The difference in magnitude between EFRs recorded for different stimulus carriers and for different stimulus levels on the CochSyn test prototype with Snap electrodes and the cEEGrid electrodes during session 1.
Gender differences in EFR magnitude | end of session 1, after 3 hours
  The difference in EFR magnitude between men and woman of the cohort recorded on the CochSyn test prototype with Snap electrodes and the cEEGrid electrodes during session 1.
Selectivity of EFR measurements | end of session 1, after 3 hours
  The difference between the EFR magnitudes of the control group and the test group for different stimulus carriers during session 1. Recordings are made on the CochSyn test prototype + Snap electrodes and differences will be assessed across the age-cohort as well as within each age group.
Age-related decline in EFR magnitude | end of session 1, after 3 hours
  The correlation strength and regression slope of the EFR magnitudes with age obtained with the CochSyn test prototype + Snap electrodes measured at different carrier frequencies and sound levels during session 1 for the test subjects with or without self-reported hearing difficulties.
Subjective hearing handicap | end of session 1, after 3 hours
  The correlation between the HHIE-s questionnaire score and the EFR magnitude at different carrier frequencies obtained with the CochSyn test prototype + Snap electrodes during session 1.
Classification accuracy scale | session 1, after 3 hours
  Classification accuracy scale of correctly assigning a subject within a specific age group to have a subjective hearing handicap (based on HHIE-s) based on their EFR magnitude.
Hearing thresholds | end of session 1, after 3 hours
  The correlation strength and regression slope of the EFR magnitude with the hearing threshold across the cohorts with and without self-reported hearing difficulties. Hearing thresholds related to standard clinical measures i.e., the pure-tone average from the audiogram with extended frequencies and distortion-product otoacoustic emission thresholds. EFR magnitudes at different carrier frequencies and sound levels during session 1 are considered.
Speech intelligibility | end of session 1, after 3 hours
  The correlation strength and regression slope of the EFR magnitude with the speech reception threshold (objective marker of speech intelligibility, Matrix sentence test) across the cohorts with and without self-reported hearing difficulties. EFR magnitudes at different carrier frequencies and sound levels during session 1 are considered.
Performance of CoNNear soundprocessing algorithm for normal audiograms | end of session 2, after 2,5 hours
  The speech reception threshold change (in dB) for subjects with low EFR magnitudes and normal audiograms that have received personalised CoNNear audio-processing to compensate for their low EFR magnitudes. The baseline situation is the speech reception threshold for unprocessed sound from session 2.
Performance of CoNNear soundprocessing algorithm for impaired audiograms | end of session 2, after 2,5 hours
  The speech reception threshold change (in dB) for subjects with low EFR magnitudes and impaired audiograms that have received personalised CoNNear audio-processing to compensate for their low EFR magnitudes. The baseline situation is the speech reception threshold for unprocessed sound from session 2 and a standard sound processing algorithm.
Sound quality rating of CoNNear soundprocessing algorithm | session 2, after 2,5 hours
  The difference in sound quality rating for the different CoNNear processing types compared to the unprocessed test material.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Verhulst, Prof., Study Director — University Ghent
Locations (1):
- UZ Gent - department of otorhinolaryngology, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No